CLINICAL TRIAL: NCT00157781
Title: Low Energy in Atrial Fibrillation AF Phase IV Study in AT/AF Population Atrial Arrhythmias Prevention and Reduction With Low Energy Atrial Antitachycardia Pacemaker
Brief Title: LEAF - Low Energy In Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 124; CP00/63 (CCPPRB Lille France); 2001/08/010 (AFSSAPS France)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Atrial Tachyarrhythmia
Keywords: Atrial Fibrillation; Atrial Tachyarrhythmia; Pacing; Electrophysiology
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Device: Medtronic AT500

SUMMARY:
The purpose of the study is to demonstrate the efficiency on AT / AF prevention and termination of a new algorithm contained in the Medtronic AT500 Antitachycardia device in patients with conventional pacemaker indications.

DETAILED DESCRIPTION:
Aim. More than 30% of patients (pts) implanted with a pacemaker are known to have atrial tachyarrhythmias (AT) despite medical treatment and about 20% of pts experience AT prior to implant. The Medtronic AT500TM is a new DDDRP pacemaker with extended memory and features designed for preventing and terminating AT. The objective of this European multi-center prospective crossover and randomized study is to evaluate efficacy of this device for decreasing AT burden, improving QOL and reducing symptoms and costs. Method. 243 pts are implanted with the AT500TM and followed at 1, 7 and 13 months after implant. All patients are selected for a dual chamber pacemaker indication plus at least two episodes of AT in the last 12 months. One month after implantation patients are randomized either to a six month therapy phase (activation of preventive and ATP pacing) or a six month observation phase (No AT prevention nor Therapy). Crossover (CO) takes place at seven months after implant and the endpoint is reached at 13 months. Symptom checklist and QOL questionnaires are completed by pts at enrollment and after the two randomization periods. At each follow-up, a Save to Disk (STD) of device-stored AT episodes is performed and hospitalization, visits and/or other examinations are reported for future cost evaluation.

ELIGIBILITY:
Inclusion Criteria:

* ACC/AHA Class I or II indication for dual chamber pacing and two symptomatic atrial fibrillation or flutter episodes in the three months prior to implant as well as ECG documentation of at least one episode in the prior year.

Exclusion Criteria:

* Patients with permanent/persistent AF, an indication for an implantable cardioverter defibrillator or class IV heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237
Dates: Start 2000-08; Study Completion 2003-11

PRIMARY OUTCOMES:
Demonstrate that AT 500 algorithms decrease AF Burden

SECONDARY OUTCOMES:
Characterize the efficiency of prevention and termination algorithms on the Quality of Life of patients
Characterize the correlation between symptoms and stored EGM's
Determine the total number of AF/AT episodes and observe the decrement of their occurrence frequency due to prevention algorithms.
Determine the number of Hospitalization, physician visits…: economical analyze
Analyze the episode onset mechanism

CONTACTS AND LOCATIONS:
Overall Officials: Kacet Salem, Prof., Principal Investigator — University Hospital, Lille; Mabo Philippe, Prof., Study Chair — CHU Rennes,France; Pisipia André, Dr., Study Chair — Hopital St Joseph - Marseille - France; Frank Robert, Dr., Study Chair — CHU Pitié-Salpétrière - Paris - France; Attuel Patrick, Dr., Study Chair — Clinique Parly 2 - le Chesnay - France; Aliot Etienne, Prof., Study Chair — CHU Nancy - France; le Heuzey Jean Yves, Prof., Study Chair — HEGP Paris - France; Davy Jean Marc, prof., Study Chair — CHU Montpellier - France; Defaye Pascal, Dr, Study Chair — CHU Grenoble - France